CLINICAL TRIAL: NCT00802945
Title: A Multicenter, Open-Label, Phase 2 Study to Evaluate the Safety and Efficacy of NKTR-102 When Given on a Q14 Day or a Q21 Day Schedule in Patients With Metastatic or Locally Advanced Breast Cancer Whose Disease Has Failed Prior Taxane-Based Treatment
Brief Title: Study to Evaluate the Safety and Efficacy of NKTR-102 in Patients With Metastatic or Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-PIR-05
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Tumor; Breast Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — etirinotecan pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NKTR-102 q14d (Experimental): NKTR-102
  Interventions: Drug: NKTR-102
- NKTR-102 q21d (Experimental): NKTR-102
  Interventions: Drug: NKTR-102

INTERVENTIONS:
Drug: NKTR-102 — NKTR-102 given on a q14 day schedule
  Arms: NKTR-102 q14d
Drug: NKTR-102 — NKTR-102 given on a q21 day schedule
  Arms: NKTR-102 q21d

SUMMARY:
This is a multicenter, open-label, two-arm, 2-stage, Phase 2 study of NKTR-102 in patients with metastatic or locally advanced breast cancer whose disease has failed prior taxane-based treatment in the metastatic setting.

Patients will be randomized 1:1 into one of two treatment arms. NKTR 102 will be administered at a dose level of 145 mg/m2 in both arms. In Arm A, NKTR-102 will be given on a q14d schedule. In Arm B, NKTR-102 will be given on a q21d schedule. Approximately 70 patients may be evaluated in this study with approximately 35 patients enrolled in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Inoperable metastatic or locally advanced breast cancer
2. No more than 2 prior chemotherapy regimens given in a metastatic or locally advanced setting and prior treatment in the metastatic setting must have included a taxane

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to Day 1 of Cycle 1
2. Patients who have had any major surgery within 4 weeks prior to Day 1 of Cycle or minor surgery within 2 weeks prior to Day 1 of Cycle 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Hannah, MD, Study Director — Nektar Therapeutics
Locations (19):
- United States (8):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - Stockton Hematology/Oncology, Stockton, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Louisville Oncology Clinical Research Program, Louisville, Kentucky
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Pharma Resource, East Providence, Rhode Island
  - University of Virginia Health System, Charlottesville, Virginia
- Belgium (5):
  - Institut Jules Bordet, Brussels
  - UZ Antwerpen, Edegem
  - De Pintelaan 1885, Ghent
  - CHU de Liege, Liège
  - GasthuisZusters Antwerpen, Wilrijk
- United Kingdom (6):
  - Clatterbridge Centre for Oncology, Bebington
  - Velindre Hospital, Cardiff
  - Beatson Oncology Center, Glasgow
  - St James University Hospital, Leed
  - Nottingham City Hospital, Nottingham
  - Weston Park Hospital, Sheffield

REFERENCES:
- [Derived] Awada A, Garcia AA, Chan S, Jerusalem GH, Coleman RE, Huizing MT, Mehdi A, O'Reilly SM, Hamm JT, Barrett-Lee PJ, Cocquyt V, Sideras K, Young DE, Zhao C, Chia YL, Hoch U, Hannah AL, Perez EA; NKTR-102 Study Group. Two schedules of etirinotecan pegol (NKTR-102) in patients with previously treated metastatic breast cancer: a randomised phase 2 study. Lancet Oncol. 2013 Nov;14(12):1216-25. doi: 10.1016/S1470-2045(13)70429-7. Epub 2013 Oct 4. PMID 24095299

RESULTS

PARTICIPANT FLOW:
Groups:
- NKTR-102 14 Day: NKTR-102: NKTR-102 given on a q14 day schedule
- NKTR-102 21 Days: NKTR-102: NKTR-102 given on a q21 day schedule
Period: Overall Study
Arm/Group | NKTR-102 14 Day | NKTR-102 21 Days
Started | 35 | 35
Completed | 0 | 0
Not Completed | 35 | 35
Not completed — Death | 27 | 23
Not completed — Terminated by sponsor | 8 | 12

BASELINE CHARACTERISTICS:
Groups:
- NKTR-102 14 Day: NKTR-102
  NKTR-102: NKTR-102 given on a q14 day schedule
- NKTR-102 21 Days: NKTR-102
  NKTR-102: NKTR-102 given on a q21 day schedule
- Total: Total of all reporting groups
Arm/Group | NKTR-102 14 Day | NKTR-102 21 Days | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 28 | 57
  >=65 years | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (12.3) | 55.8 (10.5) | 54.5 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 69
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 14 | 12 | 26
  United States | 7 | 10 | 17
  United Kingdom | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | NKTR-102 14 Day | NKTR-102 21 Days
Number analyzed (Participants) | 35 | 35
percentage of subjects | 28.6 [14.6 to 46.3] | 35 [14.6 to 46.3]

2. Secondary Outcome: Kaplan Meier Estimate of Progression-Free Survival (PFS)
Description: Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions", or similar definition as accurate and appropriate.
Time Frame: Up to 2 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 14 Day | NKTR-102 21 Days
Number analyzed (Participants) | 35 | 35
Months | 3.3 [2.6 to 5.7] | 5.6 [1.8 to 6.2]

3. Secondary Outcome: Kaplan Meier Estimate of Overall Survival (OS)
Description: OS was calculated as the time from the date of first study drug administration until death from any cause. Subjects alive at the time of analysis were censored at the time they were last known alive. OS was analyzed for the ITT population.
Time Frame: Up to 2 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 14 Day | NKTR-102 21 Days
Number analyzed (Participants) | 35 | 35
Months | 8.8 [5.4 to 15.0] | 13.1 [9.2 to 19.2]

4. Secondary Outcome: Kaplan Meier Estimate of 6-month Survival
Description: Six-month survival (i.e., overall survival proportion at 6 months) was estimated using Kaplan Meier method. The analyses were performed in the ITT population.
Time Frame: From Cycle 1 Day 1 to the end of 6 months.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | NKTR-102 14 Day | NKTR-102 21 Days
Number analyzed (Participants) | 35 | 35
percentage of subjects | 57.1 [39.3 to 71.5] | 82.9 [65.8 to 91.9]

5. Secondary Outcome: Kaplan Meier Estimate of 1-year Survival
Description: One year survival (i.e., overall survival proportion at 12 months) was estimated using Kaplan Meier method. The analyses were performed in the ITT population.
Time Frame: From Cycle 1 Day 1 to the end of 12 months.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | NKTR-102 14 Day | NKTR-102 21 Days
Number analyzed (Participants) | 35 | 35
percentage of subjects | 42.9 [26.4 to 58.3] | 51.4 [34.0 to 66.4]

6. Secondary Outcome: Percent of Patients With Treatment-Emergent Adverse Events (TEAE): NCI-CTCAE Grade 3 or Higher With Incidence Rate ≥ 2% in Either Treatment Group
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not thought to be related to the investigational product. TEAE was any event not present before exposure to the study drug or any event already present that worsened in either intensity or frequency after exposure to the study drug. All AEs were assessed for severity using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 3.0. If a particular AE was not listed in the NCI CTCAE Version 3.0, the following criteria were used: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life threatening or disabling; Grade 5 = Death.
Time Frame: Up to 2 years.
Measure: Number; unit: percentage of subjects
Arm/Group | NKTR-102 14 Day | NKTR-102 21 Days
Number analyzed (Participants) | 35 | 35
percentage of subjects
  Percentage of Patient with at Least 1 TEAE | 68.6 | 54.3
  Diarrhoea | 20.0 | 22.9
  Nausea | 5.7 | 2.9
  Fatigue | 14.3 | 8.6
  Vomiting | 8.6 | 5.7
  Decreased appetite | 2.9 | 0
  Abdominal pain | 2.9 | 0
  Dehydration | 8.6 | 11.4
  Neutropenia | 11.4 | 11.4
  Anaemia | 2.9 | 2.9
  Dyspnoea | 2.9 | 0
  Disease progression | 14.3 | 8.6
  Lethargy | 2.9 | 0
  Dizziness | 2.9 | 2.9

ADVERSE EVENTS:
Time Frame: From the time of informed consent to the last study visit (30 days after the last infusion of study drug), up to 2 years.
Arm/Group | NKTR-102 14 Day | NKTR-102 21 Days
All-Cause Mortality (participants affected / at risk) | 27/35 | 23/35
Serious Adverse Events (participants affected / at risk) | 18/35 | 15/35
Other Adverse Events (participants affected / at risk) | 35/35 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NKTR-102 14 Day (N=35) | NKTR-102 21 Days (N=35)
Lymphoedema (Vascular disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Disease Progression (General disorders) | 4 | 3
Fatigue (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 0
Blood Pressure Decreased (Investigations) | 0 | 1
ECG Signs Of Myocardial Ischaemia (Investigations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Monoplegia (Nervous system disorders) | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Vision Blurred (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Ileitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Neutropenic Sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Septic Shock (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-102 14 Day (N=35) | NKTR-102 21 Days (N=35)
Hypotension (Vascular disorders) | 3 (3) | 1 (1)
Weight decreased (Investigations) | 3 (4) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 5 (9) | 7 (19)
Dizziness (Nervous system disorders) | 2 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 3 (4) | 4 (5)
Headache (Nervous system disorders) | 4 (4) | 4 (5)
Lethargy (Nervous system disorders) | 3 (6) | 5 (6)
Paraesthesia (Nervous system disorders) | 3 (3) | 1 (1)
Vision blurred (Eye disorders) | 8 (11) | 6 (11)
Asthenia (General disorders) | 4 (7) | 2 (2)
Fatigue (General disorders) | 15 (55) | 18 (31)
Oedema peripheral (General disorders) | 4 (4) | 2 (2)
Pain (General disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 4 (5) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 7 (9) | 8 (11)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 4 (5)
Constipation (Gastrointestinal disorders) | 14 (21) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 24 (58) | 27 (61)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 24 (33) | 26 (36)
Vomiting (Gastrointestinal disorders) | 18 (33) | 14 (18)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (8) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 14 (15) | 12 (15)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (7) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 2 (3)

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of subjects analyzed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.